CLINICAL TRIAL: NCT07016932
Title: Independent Life Support Program; Determination of the Effectiveness of Menstruation Management Training Given With Mobile Application (Independent I Can) in Female Adolescents With Mild Intellectual Disabilities
Brief Title: Menstrual Management Using a Mobile Application in Adolescent Girls With Mild Intellectual Disabilities
Acronym: Independent
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Hacer ALAN DİKMEN, Assos. Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/288; 323S198 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-05-15; First posted 2025-06-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Mother; Menstrual Hygiene Management; Hand Hygiene; Intellectual Disability, Mild
Keywords: mild intellectual disability; adolescent; mother; menstruation management; hand hygiene
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: After randomization, female adolescents with mild intellectual disabilities will be trained with the mobile application (I Can Do It Independently) in addition to routine education. The mobile application will be introduced to the mothers of the female adolescents and installed on their phones. Then, the mothers will be asked to create a "user name and password" and will be registered to the mobile education application. In the meantime, the mothers will be told again how to use the mobile training application. I can do it independently was developed by the researchers. During the mobile application development process, suggestions were received from experts and the mobile application was finalized. Mild female adolescents in the experimental group were required to watch hand hygiene and menstruation management videos on the mobile application every day and play the games that followed. The researcher will call the mothers twice a week to inquire about their mobile application usage. T
Who Masked: Participant, Outcomes Assessor
Masking Description: The mild female adolescents in the experimental group are required to log in to the mobile application every day, watch the hand hygiene and menstruation management videos, and play the games that follow. The mothers will be called twice a week by the researcher to ask about their mobile application usage. Therefore, researcher blinding will not be performed. The data for the study is collected by an interviewer.
  In the study, a single blinding method in which the participants are blinded will be used. In order to prevent detection bias, data collection forms will be collected by the interviewer who has no knowledge about the research groups. In order to prevent reporting bias, the data obtained from the research will be coded as A and B by an independent researcher and transferred to the SPSS programme, and the analysis of the data coded in terms of groups will be carried out by an independent statistical expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application group (Experimental): After randomization, female adolescents with mild intellectual disabilities will be trained with the mobile application (I Can Do It Independently) in addition to routine education. The mobile application will be introduced to the mothers of the girl adolescents and installed on their phones. Then, the mothers will be asked to create a "user name and password" and will be registered to the mobile education application. In the meantime, the mothers will be told again how to use the mobile education application. I Can Do It Independently was developed by the researchers. During the mobile application development process, suggestions were received from experts and the mobile application was finalized. Mild level female adolescents in the experimental group were required to enter the mobile application every day, watch hand hygiene and menstruation management videos and play the games that followed. Mothers will be called twice a week by the researcher and their mobile application usage
  Interventions: Behavioral: Education with mobile application
- Control group (No Intervention): The routine education program will be applied to the mildly mentally retarded female adolescents assigned to the control group, and after the data are collected, the mothers and female adolescents in the control group will also be trained by the researchers with the mobile application.

INTERVENTIONS:
Behavioral: Education with mobile application — The "I Can Do It Independently" mobile application developed by the researchers includes two training videos on hand hygiene and menstruation management. Adolescents will be asked to play the games related to the training after watching the training videos. Thus, it is aimed for the participant to reinforce the training. The mobile application was developed by a multidisciplinary team of special education, nurse, midwife and software engineering academicians specifically for female adolescents with mild intellectual disabilities. Adolescents in the intervention group will be asked to use the mobile application for approximately 30 minutes every day. (https://play.google.com/store/apps/details?id=com.hookey.bagimsizyapabilirim&pcampaignid=web_share)
  Arms: Mobile application group

SUMMARY:
In the study conducted to determine the effectiveness of menstruation management training given with a mobile application (Bağımsız Yapabilirim) in female adolescents with mild intellectual disabilities in the independent living support program, the effect of the developed mobile application on hand hygiene and pad change will be determined. The research is a randomized controlled study.

DETAILED DESCRIPTION:
When the existing literature is examined, it is seen that there are limited number of studies on menstruation management education. In the studies, menstrual hygiene education was given to mentally disabled adolescent girls in small groups with model dolls or videos on social media that were not prepared by experts. Although these studies show that menstrual hygiene education given to mentally disabled students is successful, they are limited to small sample groups. For adolescent girls with intellectual disabilities, the onset of menstruation affects their independence and creates additional concerns for mothers at home, at school and in other settings. In studies conducted with mothers of adolescent girls with intellectual disabilities, mothers reported that they worried about their daughters' inability to understand menstruation, inability to change pads or dispose of them in the trash can appropriately, inability to pay attention to privacy during these special days, and that they did not send their daughters to school because they thought that they could not manage the menstruation process. Mothers' worries and fears during this process cause adolescent girls with intellectual disabilities to spend approximately one week at home every month, preventing them from socializing, negatively affecting their academic skills, further slowing their developmental processes and making it difficult for them to get used to independent life. In addition, studies show that the quality of life of both mothers and girls decreases significantly due to poor management of the menstruation process.

The main aim of this study was to determine the effectiveness of menstruation management training given to female adolescents with mild intellectual disabilities using a mobile application (Bağımsız Yapabilirim).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild intellectual disability
* Menstrual cycle has started and menstruation is regular
* Primary caregivers are mothers
* Toilet-trained
* Has the ability to stick an adhesive object to a surface and remove it from the surface
* Have the ability to dress and undress
* Have the ability to follow simple instructions
* Adolescent girls and their mothers who have the ability to recognize the materials to be used will be included in the study.

Exclusion Criteria:

* Not willing to use the mobile application at any stage of the study
* Participated in a different training on menstruation management while the research was ongoing
* Not completing the education process
* Not completing the data collection forms
* Mentally disabled adolescent girls with moderate, severe and very severe intellectual disabilities and their mothers will be excluded from the study.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 82 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Form for Mothers and Female Adolescents with Intellectual Disabilities | 1st Time: Day 1
  This form was developed through a literature review to be used in both "analysis" and "design" phases of the study. The form consists of two sections to determine the socio-demographic characteristics of mothers and daughters and the menstrual characteristics of the mentally disabled female adolescent. In the first part of the form in which socio-demographic characteristics were evaluated, there were 17 questions such as the age of the mother and daughter, education and employment status of the mother, while in the second part of the form in which menstrual characteristics of the mentally disabled female adolescent were evaluated, there were 11 questions about menstruation period and hygiene such as whether menarche started or not, whether menstrual cycle was regular or not, whether the mother gave education to her daughter about menstrual period and pad change or not.

SECONDARY OUTCOMES:
Hand Hygiene Skill Performance Recording Chart | 1st Time: Day 1, 2nd Time: Day 30, 3rd Time: Day 90, 4th Time: Day 240
  This form was created according to the hand washing guide of the Ministry of Health to be used in the "implementation" phase of the study according to the ADDIE learning design model and in the experimental and control groups in the final phase of the study. The form includes 10 statements created in accordance with the hand hygiene steps in order to measure the hand hygiene skills of female adolescents.

OTHER OUTCOMES:
Menstrual Care (Using Pads) Skill Performance Record Chart | 1st Time: Day 1, 2nd Time: Day 30, 3rd Time: Day 90, 4th Time: Day 240
  This form was created through a literature review to be used in the "implementation" phase of the study according to the ADDIE learning design model and in the experimental and control groups in the final phase of the study. The form includes 17 statements created in accordance with the steps of changing pads in order to measure the menstrual care (pad change) skills of female adolescents. This form will be filled out by the mothers of female adolescents with intellectual disabilities four times in total: before the application, at the end of the first, third and eighth month after the girl started using the mobile application.
Mobile Application Usability Scale | 1st Time: Day 240
  The Mobile Application Usability Scale was developed to evaluate the usability of a mobile application. It is a scale consisting of 10 factors with 4 items in each factor and 40 items in total. The scale ranges from 1 to 7 (1: Strongly Disagree, 2: Disagree, 3: Somewhat Disagree, 4: Undecided, 5: Somewhat Agree, 6: Agree, 7: Strongly Agree). There are no items that need to be reverse coded.
Mobile Application Willingness to Use Scale | 1st Time: Day 240
  To measure the willingness to use a mobile application by users. The scale, which consists of a single factor and 6 items, ranges from 1 to 7 (1: Strongly Disagree, 2: Disagree, 3: Somewhat Disagree, 4: Undecided, 5: Somewhat Agree, 6: Agree, 7: Strongly Agree) Likert-type scale. There are no items that need to be reverse coded in the scale.
Mobile Application Usage Loyalty Scale | 1st Time: Day 240
  To determine users' usage loyalty for a mobile application. The scale, which consists of a single factor and 5 items, ranges from 1 to 7 (1: Strongly Disagree, 2: Disagree, 3: Somewhat Disagree, 4: Undecided, 5: Somewhat Agree, 6: Agree, 7: Strongly Agree). There are no items that need to be reverse coded.
Visual Analog Scale (VAS)-Satisfaction | 1st Time: Day 240
  VAS- satisfaction is a 10 cm long instrument. On the left end of the scale, 0=not satisfied at all and 10=very satisfied on the right end. A high score on the scale indicates a high level of satisfaction with menstruation management education, while a score of 0 indicates no satisfaction with menstruation management education.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Dikmen, Assoc. Prof., Study Director — Selcuk University
Locations (1):
- Selçuklu Özel Eğitim Meslek Okulu, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Güler, Ç. 2019. "A structural equation model to examine mobile application usability and use." Bilişim Teknolojileri Dergisi, 12(3), 169-181.
- [Result] Genç, Z., Masalimova, A., Platonova, R., Sizova, Z., Popova, O. 2019. "Analysis of documents published in scopus database on special education learning through mobile learning: A content analysis". International Journal of Emerging Technologies in Learning (IJET), 14(22), 192-203.
- [Result] Bakır, D., Demirli, C. 2020. "Investigation of the impact of self-compassion and family support perception on parenting stress in parents who have children with learning disability, autism spectrum disorder and mental disability". Humanistic Perspective, 2 (3), 271-282 .
- [Result] Açar, D., Dilbilir, Y., Demiralp, C. 2022. "Özel eğitim öğretmenlerinin zihinsel yetersizliği olan çocukların eğitimi sürecindeki görüşlerinin incelenmesi". Abant İzzet Baysal Üniversitesi Eğitim Fakültesi Dergisi, 22(3), 1295-1312.
- See also: link to the mobile app — https://play.google.com/store/apps/details?id=com.hookey.bagimsizyapabilirim&pcampaignid=web_share